CLINICAL TRIAL: NCT02897934
Title: Continuous Wound Infiltration and 23 Hour Discharge Following Major Breast Cancer Surgery
Brief Title: CWI and Discharge After Breast Cancer Surgery
Status: Completed | Type: Observational
Sponsor: University College Cork (Other)
Responsible Party: Principal Investigator, Brian Declan O'Donnell, Consultant Anaesthetist and Clinical Senior Lecturer, University College Cork
Other Study IDs: ECM4(h)031115
Record Dates: First submitted 2016-08-31; First posted 2016-09-13 (Estimated); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Breast Cancer; Pain
MeSH Terms: conditions — Breast Neoplasms; Pain | interventions — Bupivacaine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Bupivacaine continuous infusion — The use of continuous wound infusion of bupivacaine
  Other Names: marcain

SUMMARY:
The objectives of this work are threefold:

1. To evaluate the analgesic efficacy of CWI in women discharged within 23 hours of major breast cancer surgery
2. To evaluate objective indices of patient recovery following anaesthesia and surgery in a 23 hour model of care
3. To evaluate patient satisfaction with their care pathway

DETAILED DESCRIPTION:
Cork University Hospital is a designated cancer centre, under the national Cancer Control Programme treating in excess of 560 new cases of breast cancer each year. Breast surgery is performed by five specialist breast surgeons, with patients accessing services from either the National Cancer Screening Programme (BreastCheck) or via referral from family physicians to the rapid access symptomatic breast assessment unit. Both acute and persistent pain following incisional breast surgery is a significant problem. In the past, it has been reported that up to 50% of women undergoing incisional breast surgery experience significant pain immediately following surgery. One in three women may develop persistent post surgical pain lasting greater than 3 months. The use of multimodal analgesic regimen to include non-steroidal anti-inflammatories, paracetamol, low dose opiates and importantly local anaesthetic techniques have seen a significant improvement in post-operative pain management following incisional breast surgery. Local anaesthetic techniques such as paravertebral blockade have become commonplace in the management of pain following major incisional breast surgery.

Current budgetary difficulties have brought increased pressures to bear upon the use and availability of hospital beds. This has resulted in a shift from an inpatient model of care to a day case model. More than 85% of all breast cancer surgery is performed as day cases (same day admission/discharge). The remainder of breast cancer surgeries require a same day admission with variable length of stay post-operatively. Pain is a significant determinant of length of post operative stay. Patients with moderate to severe pain are less independent, require assistance with basic care, consume opiate analgesics, suffer opiate-related side effects, are less compliant with post-operative physiotherapy and consume more healthcare resources than patients with mild or no pain. Therefore the design and implementation of an effective pain management strategy for women undergoing major incisional breast surgery is an essential component to the overall perioperative patient care pathway.

Since 2010, patients undergoing major incisional breast surgery through BreastCheck at Cork University Hospital have received a multimodal analgesic regimen during and following surgery which is based upon the use of local anaesthetic continuous wound infiltration (CWI). The efficacy of CWI following mastectomy has been found to be equivalent to the gold standard paravertebral block. Similarly, the efficacy of CWI in women undergoing axillary lymph node dissection has previously been demonstrated. The clinical experience of women undergoing mastectomy with axillary clearance or sentinel node surgery suggest equivalence between paravertebral analgesia and CWI.

Since January 2013, women undergoing major breast cancer surgery at Cork University Hospital have been enrolled in a prospective cohort study to evaluate the efficacy of an enhanced perioperative pathway. Elements of this pathway include improved process flow with the establishment of dedicated preoperative assessment and preadmission clinics, day of surgery hospital admission and an admission lounge adjacent to the operating theatres, standardised anaesthesia, analgesia and surgical protocols, goal based immediate post-operative recovery, early independent ambulation and enteral nutrition, active discharge planning and early assessment of hospital discharge readiness. Although women following major breast cancer surgery achieve hospital discharge readiness scores early, the length of hospital stay is determined by institutional and individual clinician convention, rather than objective assessment of home readiness.

Parallel to work on the enhanced perioperative pathway, clinicians at Cork University Hospital have devised APP based technology which will be integrated into the perioperative pathway. Prior to surgery, the APPs will provide both clinician and user generated educational material relating to first person perspective on perioperative experiences. In the post-operative phase, the technology will enable clinicians to monitor and interact with patients remotely, thereby facilitating early hospital discharge. The technology will also enable patients to communicate anonymously with each other, generating contemporaneous communities of recovery.

The objectives of this work are threefold:

to identify, characterise and manage barriers to safe discharge within 23 hours of major breast cancer surgery; to evaluate the feasibility of discharging a select cohort of patients at 23 hours following major breast cancer surgery with indwelling CWI as the mainstay of post operative analgesia to evaluate the analgesic efficacy of CWI in women discharged within 23 hours of major breast cancer surgery

Primary Endpoint:

The analgesic efficacy and safety of CWI in women discharged home within 23 hours of major breast cancer surgery as assessed by patient reported pain scores 24 and 48 hours discharge, and surveillance to detect adverse events associated with CWI use.

Secondary Endpoints:

Quality of recovery at 24 & 48 hours (QoR 40) Analgesic Consumption at 24 & 48 hours Wound drain output at 24 & 48 hours Patient Satisfaction Score

Preoperatively, patients will be screened at the preassessment clinic and their suitability for 23 hour discharge will be assessed according to institutional norms. The patients will receive preoperative, nurse delivered education regarding wound care and wound drain management. A mutually agreed discharge plan will be designed between the patient and the multidisciplinary team. The patient will receive their perioperative technology device and become familiar with the educational and communications functionality contained within.

On the day of surgery patients will be admitted to the operating theatre day of surgery area (DOSA). In DOSA they will have the opportunity to meet the perioperative team again and ask any outstanding questions. They will then change into a theatre gown and enter the operating theatre.

This patient cohort will receive standard propofol TIVA (T4 TIVA protocol attached). With standard monitoring in place (pulse oximetry, electrocardiography, non-invasive arterial blood pressure and inspired and end- tidal partial pressures of O2 and CO2), patients will receive preinduction Fentanyl 100mcg and Midazolam 2mg. Entropy processed frontal lobe EEG monitoring will be attached. Anaesthesia will be induced with propofol target controlled infusion (Marsh Algorithm; 4-6mcg/ml dose range using 2% Propofol) and the lungs will be assist ventilated in 65% oxygen/air mixture. Airway and intraoperative fluid management is entirely at the discretion of the responsible consultant anaesthetist.

Intraoperative analgesia:

Patients will receive Diclofenac 75mg and Paracetamol 1g during surgery. Administration of intraoperative morphine up to 0.1mg/kg will be at the discretion of the consultant anaesthetist. All patients will be given PONV prophylaxis with ondansetron 4mg and dexamethasone 8mg intraoperatively.

Wound soakage with 40ml of 0.25% bupivacaine with 1:200,000 adrenaline will be performed by the surgeon, allowing a minimum of 3 minute soakage time prior to wound closure. Two multiple port catheters will be placed by the surgeon, one directed towards the chest wound and the other towards the axillary wound. These catheters will then be connected up to the prefilled INFUSOR single use pump delivering 5 ml/hr of 0.25% bupivacaine.

Postoperatively, all patients will be transferred from theatre to the post anaesthesia care unit (PACU) where they will remain until PACU discharge criteria are met. In the PACU, if patients experience pain, 10 ml of 2% Lidocaine will be administered through the catheters in CWI in the first instance. Morphine 2mg IV PRN may be administered as rescue analgesia if required thereafter. Patients may be administered additional antiemetics (Ondansetron) in the PACU.

Following transfer to the ward, all patients will receive a standard analgesic regimen of Diclofenac sodium, 75 mg PO 12 hourly/ PRN and Paracetamol, 1 g PO/PR, 6 hourly /PRN, and Oxycodone (Oxynorm) 10mg 4 hourly /PRN.

While in hospital, data in relation to patient recovery, pain and complications will be recorded using Cork University Hospital's perioperative pathway clinical data sheet. Following discharge, postoperative data will be collected using a bespoke android app specifically designed to capture outcome measures on the first and second post operative days. The app gathers anonymised data in relation to pain (slide-rule page analogous to the visual analogue score), quality of recovery (QoR40 Score), wound drain output in millilitres and patient satisfaction on a likert-type scale. Data will be collected following discharge on the first and second postoperative days. Participants will be encouraged to provide free-text feedback in relation to their healthcare experience. Any adverse events will be monitored, recorded and treated appropriately.

Summary data with respect to the primary and secondary endpoints will be presented. Where appropriate, 95% confidence intervals will be calculated.

ELIGIBILITY:
Inclusion Criteria:

Women undergoing any one of:

mastectomy mastectomy with axillary lymph node clearance mastectomy with axillary lymph node sampling

Exclusion Criteria:

Refusal to participate; Allergy to Bupivacaine; Pre-existing pain conditions; Regular use of opioid analgesia; Pregnancy; Uncontrolled Diabetes; Uncontrolled Thyroid disorder; Severe cardiac, renal or hepatic disease ; Bilateral surgery; Planned discharge >23 hours; Travel time from the admitting hospital >45 minutes; Absence of intellectual capacity to consent

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women undergoing mastectomy and mastectomy with axillary surgery.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2016-08; Primary Completion 2018-01-01 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Pain | 24 hours, 48 hours
  Pain will be recorded at at 24 and 48 hours using a slide-rule page on bespoke Android App. Pain will be recorded in a manner analogous to a visual analog scale 0 = No pain, 100 = Worst imaginable pain. Participants will be prompted on the first and second postoperative days to score their worst level of pain.

SECONDARY OUTCOMES:
Quality of recovery at 24 & 48 hours (QoR 40) | 24 hours, 48 hours
  The quality of postoperative recovery from surgery and anaesthesia will be scored on the first and second postoperative day using the validated QoR 40 score. These metrics will be recorded on a bespoke Android App.
Analgesic Consumption at 24 & 48 hours | 24 hours, 48 hours
  The quantity of analgesics consumed on the first and second post operative day will be recorded, on a bespoke Android App.
Wound drain output at 24 & 48 hours | 24 hours, 48 hours
  Wound drain serous fluid output will be measured as is usual by the patient. These metrics will be recorded on a bespoke Android App.
patient satisfaction | 48 hours
  Patient satisfaction with their perioperative experience will be measured on a likert-type scale using a bespoke android app.

CONTACTS AND LOCATIONS:
Overall Officials: Brian O'Donnell, MD, Principal Investigator — Cork University Hospital
Locations (1):
- Brian O'Donnell, Cork, Ireland

IPD SHARING:
Plan to Share IPD: No
Only pooled data will be shared/reported